CLINICAL TRIAL: NCT05937204
Title: Nursing Teaching Scheme to Improve Remedial Compliance and Alleviate Symptoms Among Patients With Gastro-esophageal Reflux Disease
Brief Title: Nursing Teaching Scheme for Patients With Gastroesophageal Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa mahmoud goumaa mahmoud, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: nursing teaching scheme - GERD
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Compliance; Symptoms
MeSH Terms: conditions — Gastroesophageal Reflux; Patient Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one group pre- test post- test (Experimental)
  Interventions: Other: Nursing Teaching

INTERVENTIONS:
Other: Nursing Teaching — A nursing teaching scheme refers to a systematic and structured plan developed by nurses to provide teaching and instruction to patients. The components of a nursing teaching scheme typically include assessing learning needs, setting learning objectives, developing teaching materials, delivering information using various teaching methods, demonstrating skills, providing written instructions, assessing learning outcomes, and conducting follow-up

SUMMARY:
The aims of the study are:

* Assess patient's level of knowledge regarding gastroesophageal reflux disease.
* Assess patient' compliance and symptoms of gastroesophageal reflux disease.
* Design and implement nursing teaching scheme for patients with gastroesophageal reflux disease.
* Evaluate the effect of nursing teaching scheme on patient' compliance and symptoms of gastroesophageal reflux disease.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is one of the most common gastrointestinal disorders, which resulting from a retrograde flow of part of the gastroduodenal contents into the esophagus. Generally, this reflux is linked to a malfunction of the lower esophageal sphincter .A recent study stated that the prevalence of GERD is 18,1- 27.8% in North America, 8,8-25,9% in Europe, 2,5-7,8% in East Asia, 8,7-33,1% in middle east, 11.6% in Australia, and 23% in South America, on the other hand according to a study in Indonesia, about 3% in Asia. Many factors may contribute to the development of the disease. Among them, there are non-modifiable factors such as age, sex or genetic factors and modifiable factors, e.g. smoking, alcohol, obesity, aspirin, non-steroidal anti-inflammatory drug (NSAID) use, pregnancy. Furthermore, spicy, sour, and fatty foods can caused a direct esophageal mucosal irritation also reduction in lower esophageal sphincter (LES) tone and gastric motility. The classical symptoms of GERD are heartburn (a retrosternal burning pain radiating up towards the throat) and acid regurgitation (the perception of stomach contents coming into the hypopharynx or mouth). Atypical symptoms may also occur (including globous, chest pain, dysphagia, cough, nausea, and throat symptoms or belching). Recurrent and chronic exposure of the esophageal epithelia to the strong acidity of the refluxed material may cause esophagitis. If untreated, the disease can lead to complications such as esophageal stricture, gastrointestinal bleeding, precancerous conditions (Barrett's Esophagus ) and esophageal adenocarcinoma .Management of GERD can involve medication use, lifestyle modification, and surgical intervention depending on the individual patient and disease severity . Lifestyle interventions commonly recommended include dietary modification, weight management, smoking cessation, and head of bed elevation while recumbent and voiding recumbence at least 3 hours postprandial. The Mediterranean diet (MD) is mainly based on the regular consumption of vegetables, legumes, cereals, fruit and nuts, and the moderate consumption of ﬁsh and seafood, balanced by a comparatively limited use of red meat and other meat products, most of them cooked with olive oil as the main source of dietary fat, together with low-to-moderate alcohol consumption This diet has also been associated with a healthy lifestyle as regular physical activity and not smoking. Emerging data indicates that appropriate eating habits e.g., healthy diets involving high intakes of fruits and whole grains such as the Mediterranean diet improves GERD symptoms. Therefore, improving diets can decrease the occurrence of GERD. The crural diaphragm is one of the main components of the esophagogastric junction and plays an important role in preventing gastroesophageal reflux. The diaphragm, as a skeletal muscle, is partially under voluntary control and its dysfunction can be improved via breathing exercises. Thus, diaphragmatic breathing training (DBT) has the potential to alleviate symptoms in patients with GERD. teaching patients to do diaphragmatic breathing exercises could reduce their gastric reflux symptoms and increase their quality of life over time. Thus, diaphragmatic breathing exercises are recommended to be used as a part of these patients' treatment programs. Patient teaching has been shown to be beneficial for a variety of diseases. Patients with gastroesophageal reflux disease have wide range of unpleasant symptoms as heartburn, regurgitation so, teaching patient strategies to alleviate symptoms is important aspect .teaching is a known predictor for increased engagement in shared decision making, improved medication and treatment adherence, higher levels of satisfaction, and even better treatment outcomes.

Operational definitions:

Nursing teaching scheme:

A nursing teaching scheme refers to a systematic and structured plan developed by nurses to provide teaching and instruction to patients. The components of a nursing teaching scheme typically include assessing learning needs, setting learning objectives, developing teaching materials, delivering information using various teaching methods, demonstrating skills, providing written instructions, assessing learning outcomes, and conducting follow-up

Remedial compliance:

Compliance is defined by the World Health Organization as "the extent to which a person's behavior - taking medication, following a diet, and/or executing lifestyle changes, corresponds with agreed recommendations from a health care provider

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of gastroesophageal reflux disease

Exclusion Criteria:

* Peptic ulcer
* Esophageal cancer
* Esophageal surgery
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Symptoms of Gastroesophageal Reflux Disease | "4Weeks"
  Gastro-esophageal Reflux Disease Questionnaire. It is composed of 6 items and uses a four-graded Likert scale (0-3) to score four positive predictors of GERD (heartburn, regurgitation, sleep disturbance due to reflux symptoms, and over the medications for reflux symptoms) and a reversed Likert scale (3-0) for two negative predictors (epigastric pain and nausea), giving a total GERD score range of 0-18. The maximum score that can be obtained is 18 divided as follows mild (0- 6), moderate (7- 12) and sever (13-18)

SECONDARY OUTCOMES:
Compliance with Medication | "4Weeks"
  Mourisky Medication Adherence Scale (MMAS) It a structured self-reported 8 closed-end items response. Each response will be scored as (zero) for "no" and (one) for "yes". The total score will be calculated and the result will be categorized into two groups; the patient whose less than 4 will be categorized as non-adherent while whose score 4-8 will be categorized as adherence

CONTACTS AND LOCATIONS:
Overall Officials: shalabia elsayed abuozead, professor, Study Chair — faculty of nursing - assiut university
Locations (1):
- Faculty of Nursing Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fox M, Gyawali CP. Dietary factors involved in GERD management. Best Pract Res Clin Gastroenterol. 2023 Feb-Mar;62-63:101826. doi: 10.1016/j.bpg.2023.101826. Epub 2023 Feb 17. PMID 37094911